CLINICAL TRIAL: NCT06578793
Title: Comparison of Catheter Ablation Combined With Ethanol Ablation of the Marshall Vein vs. Catheter Ablation Alone in Persistent Atrial Fibrillation With Heart Failure: A Multicenter Randomized Controlled Study
Brief Title: Comparison of Catheter Plus Marshall Vein Ablation vs. Catheter Ablation Alone in Persistent AF With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Xuping, Chief Physician, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYSY_CAB_MVA_2024_001
Record Dates: First submitted 2024-08-22; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation, Persistent; Heart Failure
Keywords: Atrial Fibrillation; Heart Failure; Catheter Ablation; Marshall Vein
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter ablation combined with Marshall vein ethanol ablation group (Experimental): Participants in this group will undergo standard catheter ablation, which involves the isolation of the pulmonary veins and may include additional ablation of other atrial areas as necessary, guided by fluoroscopy and/or 3D electroanatomical mapping. In addition to the standard ablation procedure, participants will receive Marshall vein ethanol ablation. This involves the injection of absolute ethanol into the Marshall vein via a specialized catheter, aiming to ablate the vein's myocardial sleeves and adjacent autonomic fibers. The ethanol ablation targets arrhythmogenic substrates and aims to enhance the efficacy of the overall ablation procedure by reducing atrial fibrillation triggers.
  This combined approach is hypothesized to improve clinical outcomes by providing a more comprehensive treatment of atrial fibrillation substrates, particularly in patients with persistent atrial fibrillation and concomitant heart failure.
  Interventions: Procedure: Catheter Ablation Combined with Marshall Vein Ethanol Ablation
- Catheter ablation alone group (Active Comparator): Participants in this group will undergo standard catheter ablation, which primarily involves the isolation of the pulmonary veins, a common trigger site for atrial fibrillation. The procedure may include additional ablation of other atrial areas based on the patient's specific arrhythmogenic substrate. The catheter ablation will be performed under fluoroscopic guidance and/or with the assistance of 3D electroanatomical mapping to ensure precision. This procedure is designed to eliminate or reduce the arrhythmogenic tissue within the atria to restore and maintain normal sinus rhythm.
  This intervention is the comparator arm in the study, representing the current standard treatment for persistent atrial fibrillation, particularly in patients with concomitant heart failure.
  Interventions: Procedure: Catheter Ablation Combined with Marshall Vein Ethanol Ablation

INTERVENTIONS:
Procedure: Catheter Ablation Combined with Marshall Vein Ethanol Ablation — This study involves two procedures. The first procedure is a combination of catheter ablation with ethanol ablation of the Marshall vein. The second procedure is catheter ablation alone. Both procedures involve standard techniques used to treat persistent atrial fibrillation, with the addition of Marshall vein ethanol ablation in the experimental group aimed at potentially improving outcomes by targeting additional arrhythmogenic substrates.
  Other Names: Catheter Ablation Alone

SUMMARY:
This multicenter, randomized controlled trial aims to compare the clinical efficacy and safety of combining catheter ablation with Marshall vein ethanol ablation versus catheter ablation alone in patients with persistent atrial fibrillation (AF) and concomitant heart failure. Persistent AF is a common arrhythmia that significantly impacts the quality of life and survival rates, especially when coexisting with heart failure. While catheter ablation is a standard treatment for AF, its effectiveness in persistent AF, particularly in patients with heart failure, remains suboptimal. The addition of Marshall vein ethanol ablation may enhance treatment outcomes by targeting arrhythmogenic substrates. This study will enroll 120 participants across three centers to evaluate whether this combined approach can reduce AF recurrence, improve heart function, and enhance patient outcomes compared to catheter ablation alone.

DETAILED DESCRIPTION:
Persistent atrial fibrillation (AF) combined with heart failure presents a significant clinical challenge due to the high rates of morbidity and mortality associated with these conditions. Catheter ablation is widely used to manage AF, but its efficacy in persistent AF, particularly in patients with heart failure, is limited. Recent advances suggest that targeting the Marshall vein with ethanol ablation may offer additional benefits by disrupting critical pathways involved in AF maintenance.

This study is designed to evaluate the efficacy of combining Marshall vein ethanol ablation with standard catheter ablation compared to catheter ablation alone in a well-defined patient population. Conducted across three centers, this randomized controlled trial will rigorously assess whether the combined approach can offer superior outcomes, including lower AF recurrence rates and improved heart function. The study's findings are expected to contribute valuable insights into optimizing treatment strategies for this high-risk patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years
2. For symptomatic patients with persistent atrial fibrillation: At least a 6-month history of atrial fibrillation; atrial fibrillation duration exceeding 7 days without spontaneous conversion to sinus rhythm; at least two episodes of persistent atrial fibrillation in the past 6 months even after rhythm conversion; poor tolerance or resistance to at least one Class I, II, or III antiarrhythmic drug
3. Diagnosed with heart failure: Echocardiogram showing left ventricular ejection fraction (LVEF) ≤40%
4. Patient willing to receive medication or surgical treatment
5. Patient willing to comply with the requirements before the study, during the study, and during follow-up and to sign an informed consent form
6. Capable of completing a 6-minute walk test
7. For women of childbearing potential, a negative pregnancy test result is required

Exclusion Criteria:

1. Presence of thrombus in the left atrium
2. Left atrial diameter greater than 65 millimeters in the parasternal long-axis view, or left atrial volume exceeding 200 milliliters as measured by MRI or CT
3. Presence of significant congenital abnormalities or medical issues, deemed by the researcher as inappropriate for participation in the study
4. Reversible causes of atrial fibrillation, such as pericarditis, thyroid disease, acute alcohol intoxication, recent major surgery, or trauma
5. Currently suffering from valvular heart disease requiring surgical intervention
6. Currently suffering from coronary artery disease requiring surgical or percutaneous intervention
7. History of atrioventricular node ablation
8. Liver failure
9. Renal failure requiring dialysis
10. Contraindicated use of appropriate anticoagulation therapy
11. Participation in other experimental drug or device studies
12. Severe pulmonary disease
13. Previous catheter ablation for atrial fibrillation in the left atrium
14. Documented thromboembolic event within the past 90 days
15. Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation/Atrial Flutter (AT/AF) Recurrence | 12 months after the procedure
  The primary outcome is the proportion of participants who remain free from clinical recurrence of atrial fibrillation (AF) or atrial flutter (AFL) at follow-up. Recurrence is defined as the absence of documented AF/AFL episodes lasting 30 seconds or more during continuous ECG monitoring over a 1-month period.
Change in NT-proBNP Levels | 12 months after the procedure
  This outcome measures the change in NT-proBNP levels, a biomarker for heart failure, from baseline to follow-up, indicating the impact of the intervention on heart failure status.
Change in Left Ventricular Ejection Fraction (LVEF) | 12 months after the procedure
  This outcome assesses the change in LVEF as measured by echocardiography, reflecting the effect of the intervention on cardiac function.
Change in 6-Minute Walk Test Distance | 12 months after the procedure
  This outcome measures the change in the distance covered during the 6-minute walk test, an indicator of functional capacity and exercise tolerance.
Change in NYHA Functional Class | 12 months after the procedure
  This outcome evaluates changes in the New York Heart Association (NYHA) functional classification, which assesses the severity of heart failure symptoms and functional limitations.

SECONDARY OUTCOMES:
Presence or Absence of Arrhythmias Within 30 Days | 30 days after the procedure
  This outcome measures whether arrhythmias related to the procedure occurred within 30 days post-intervention.
Presence or Absence of Chest Tightness Within 30 Days | 30 days after the procedure
  This outcome measures whether chest tightness related to the procedure occurred within 30 days post-intervention.
Presence or Absence of Palpitations Within 30 Days | 30 days after the procedure
  This outcome measures whether palpitations related to the procedure occurred within 30 days post-intervention.
Presence or Absence of Bleeding Within 30 Days | 30 days after the procedure
  This outcome measures whether bleeding related to the procedure occurred within 30 days post-intervention.
Presence or Absence of Mortality Within 30 Days | 30 days after the procedure
  This outcome measures whether mortality related to the procedure occurred within 30 days post-intervention.
Atrial Fibrillation Burden at 6 Months | 6 months after the procedure
  This outcome assesses the percentage of time that patients experience atrial fibrillation (AF) during continuous monitoring 6 months post-intervention.
Atrial Fibrillation Burden at 12 Months | 12 months after the procedure
  This outcome assesses the percentage of time that patients experience atrial fibrillation (AF) during continuous monitoring 12 months post-intervention.
Total Number of Procedures Performed | During the procedure(s)
  This outcome measures the total number of procedures performed during the intervention.
Total Radiofrequency Ablation Time for the First Procedure | During the first procedure
  This outcome measures the total radiofrequency ablation time during the first procedure.
Total Radiofrequency Ablation Time for the Second Procedure (if applicable) | During the second procedure
  This outcome measures the total radiofrequency ablation time during the second procedure, if applicable.
Total Area of Left Atrial (LA) Tissue Ablated | During the procedure(s)
  This outcome measures the total area of left atrial (LA) tissue ablated during the procedure(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study with other researchers. The data will be used exclusively by the research team for the purposes of this study and will not be made available to third parties.